CLINICAL TRIAL: NCT03849729
Title: Effectiveness and Tolerability of Phentermine in the Reduction of Intrahepatic Fat Infiltration, Adipose Tissue and Postoperative Complications in Patients Under Bariatric Surgery
Brief Title: Effectiveness and Tolerability of Phentermine in Patients Under Bariatric Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Juarez de Mexico (Other Government)
Responsible Party: Principal Investigator, ELIZABETH PEREZ CRUZ, Principal Investigator. MD. MSc, Hospital Juarez de Mexico
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HJM0367/17-IQF
Record Dates: First submitted 2019-01-02; First posted 2019-02-21 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Obesity; Morbid Obesity; Bariatric Surgery; Non-alcoholic Fatty Liver; Weight Loss
Keywords: Obesity; Obesity treatment; Non-alcoholic Fatty Liver; Weight Loss
MeSH Terms: conditions — Obesity; Obesity, Morbid; Non-alcoholic Fatty Liver Disease; Weight Loss | interventions — Phentermine

STUDY DESIGN:
Intervention Model Description: Experimental, analytic, comparative, prospective, longitudinal and double-blinded study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phentermine (Active Comparator): Low-calorie diet + Phentermine Capsules 15 mg po by 6 weeks, one time a day before bariatric surgery.
  Interventions: Drug: Phentermine
- Placebo (Placebo Comparator): Low-calorie diet + Placebo Capsules po by 6 weeks, one time a day before bariatric surgery.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Phentermine — This is a randomized, control trial to investigate the effect and safety of Phentermine in patients with obesity who need a bariatric surgery (BMI >35 kg/m2 with comorbidities or BMI > 40 kg/m2).
  Other Names: Terfamex
  Arms: Phentermine
Other: Placebo — his is a randomized, control trial to investigate the effect and safety of Phentermine in patients with obesity who need a bariatric surgery (BMI >35 kg/m2 with comorbidities or BMI > 40 kg/m2).
  Arms: Placebo

SUMMARY:
Surgical management of Morbid Obesity is increasingly frequent. A low-calorie diet is recommended with the main goal of reducing intrahepatic fat infiltration, fat tissue and making easier the surgery. Information the use pharmacological interventions during the preoperative period in this population are rare.

DETAILED DESCRIPTION:
This is a randomized, control trial to investigate the effect and safety of Phentermine in patients with obesity who need a bariatric surgery (BMI >35 kg/m2 with comorbidities or BMI > 40 kg/m2).

Screening will be made to select eligible participants before intervention. Participants were randomly assigned to one of two groups (low-calorie diet + phentermine 15 mg or low-calorie diet + placebo) for therapies during 6 weeks. Anthropometric measurements (weight, body composition, body mass index and waist-hip index), serum metabolic profile (glucose, total cholesterol, HDL-c, LDL-c, triglycerides, and HOMA-IR) markers of inflammation (IL-1, IL-6 and PCR) and hepatic ultrasound will be measured 2 times for each participant. Surgical complications (anastomosis filtration, intestinal obstruction or stenosis, need to perform open surgery and mortality) will be evaluated. Adverse events associated with phentermine (blood pressure, cardiac frequency, headache, gastrointestinal symptoms, euphoria, anxiety and insomnia) will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Women and men
* >18 years and <55 years old.
* Diagnosis of obesity grade II with comorbidities
* Diagnosis of obesity grade III with or without comorbidities
* Approved to bariatric surgery by an interdisciplinary committee
* Having signed the Informed consent form

Exclusion Criteria:

* Use of addictive substances

  * Inability or lack of understanding to achieve lifestyle and behaviour changes
  * Mental disease
  * Severe Pulmonary disease
  * Giant Hiatal hernia, gastric or duodenal ulcer
  * Unstable coronary artery disease
  * Portal hypertension or esophageal varices
  * Surgical or anesthetic high risk

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with Intrahepatic fat | Change from baseline after 6 weeks treatment based on hepatic ultrasound.
  Intrahepatic fat semi-qualitative asessment: mild(<20%), moderate (20-30%), severe (>30%)
Fat tissue | change from baseline after 6 weeks treatment based on body composition by bioimpedance
  Fat tissue: fat mass in Kilograms and percentage

SECONDARY OUTCOMES:
Metabolic profile | Change from baseline after 6 weeks treatment based on glucose, total cholesterol, HDL-c, LDL-c, triglycerides, and HOMA-IR.
  Changes in serum metabolic profile: mg/dL
Markers of inflammation | Change from baseline after 6 weeks treatment based on IL-1, IL-6 and PCR
  Changes in serum markers of inflammation: pg/mL
Surgical complications | Surgical complications during hospitalization and up to 30 days after surgery 1) dehiscence of anastomosis, 2) intestinal obstruction, 3) intestinal stenosis
  Prevalence of surgical complications (yes or no): 1) dehiscence of anastomosis, 2) intestinal obstruction, 3) intestinal stenosis
Adverse events associated with phentermine | Adverse events during and the end of 6-8 weeks of phentermine (blood pressure, cardiac frequency, headache, gastrointestinal symptoms, euphoria, anxiety and insomnia) associated with phentermine.
  Determine the frequency and severity of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Pérez-Cruz, MD, Principal Investigator — Hospital Juárez de México
Locations (1):
- Hospital Juárez de México, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No